CLINICAL TRIAL: NCT06478147
Title: Effect of a Novel Protein Ingredient Combined With Oral Nutritional Supplement on Appetite in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Principal Investigator, Katy Horner, Lecturer in Sport and Exercise Science, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LS-22-64-Horner#2
Record Dates: First submitted 2023-11-23; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Aging; Appetite Loss; Undernutrition
Keywords: Appetite; Poor Appetite; Ageing; Whey protein hydrolysate; Visual analogue scale; Energy intake; Ghrelin; Oral Nutritional Supplement; Dairy
MeSH Terms: conditions — Anorexia; Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
  All participants undertake all three experimental conditions in a random order.
Who Masked: Participant, Investigator
Masking Description: Out of three treatments, one of the investigators is blinded for all treatments while the other is not blinded.
  The participant is fully blinded, i.e. treatments will be served in generic containers for Oral Nutritional Supplement (unlabelled) and vanilla-flavoured.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Nutritional Supplement (Placebo Comparator): 125 mL of commercially available of Oral Nutritional Supplement, a liquid food product containing vitamins, minerals, protein, fats and carbohydrates. 125 mL of product provides 37.0 g of carbohydrates, 11.6 g of fats, 12.0 g of proteins, vitamins and minerals.
  Interventions: Dietary Supplement: Oral Nutritional Supplement
- Oral Nutritional Supplement + Whey Protein Hydrolysate (Experimental): 2,2 grams of whey protein hydrolysate dissolved in 125 mL of commercially available of Oral Nutritional Supplement
  Interventions: Dietary Supplement: Oral Nutritional Supplement + Whey Protein Hydrolysate
- Whey Protein Hydrolysate (Active Comparator): 2,2 grams of whey protein hydrolysate dissolved in 125 mL of water
  Interventions: Dietary Supplement: Whey Protein Hydrolysate + still water

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplement — Commercially available Oral Nutritional Supplement alone consumed 90 minutes prior to an ad libitum breakfast
  Arms: Oral Nutritional Supplement
Dietary Supplement: Oral Nutritional Supplement + Whey Protein Hydrolysate — Whey Protein Hydrolysate dissolved in an Oral Nutritional Supplement consumed 90 minutes prior to an ad libitum breakfast
  Arms: Oral Nutritional Supplement + Whey Protein Hydrolysate
Dietary Supplement: Whey Protein Hydrolysate + still water — Whey Protein Hydrolysate dissolved in still water consumed 90 minutes prior to an ad libitum breakfast
  Arms: Whey Protein Hydrolysate

SUMMARY:
Reduced appetite can occur with ageing and is linked to a higher risk of undernutrition, poorer physical function and becoming frail. Strategies to increase appetite are needed to improve healthy ageing. This study follows on from previous work which has found a novel ingredient in whey protein (derived from whole milk) that may help to increase appetite and energy intake. This study will compare the effects of the ingredient added to an oral nutritional supplement (ONS) versus the ONS alone versus the ingredient dissolved in water on appetite in older adults. By studying this nutrition supplement in older adults, this will help to provide greater information on possible nutrition strategies to improve healthy ageing.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling,
* Age 60+ years
* Poor appetite (Simplified Nutritional Appetite Questionnaire (SNAQ) score </=14, answer a, b or c to Q.1 on SNAQ or answer b, c, or d to CES-D question regarding poor appetite in the past week)
* BMI 20-25kg/m2

Exclusion Criteria:

* Current medical condition or medication known to impact appetite or energy intake
* Other medical condition that would impact study participation and outcomes, as judged by the study investigator.
* Heavy smoker (>10/day)
* Inability to come to study centre
* Currently participating in another intervention study
* Lacking informed consent
* Allergic to or unwilling to consume any of the study test foods
* Loss of taste or smell associated with COVID-19
* Unable to walk across a room

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-06-29 (Estimated)

PRIMARY OUTCOMES:
Pre-meal and changes in Hunger | 9.5 hours: fast (pre-ONS), pre-breakfast: 90 (post-ONS), 60, 30 and 0 min; post-breakfast: 0 and 180 min (pre-lunch); post-lunch: 0 and 90 min (pre-ONS); 0 min post-ONS; estimated 120 min. post-ONS (pre-dinner); 0 min. post-dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used to assess hunger, at ten (10) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Hunger is directly obtained from its VAS rating. Changes between fast and post-meal, mean and AUC values will be calculated.
Energy Intake (EI) from an ad libitum breakfast meal (kilocalories) | Measures taken immediately following the ad libitum test meal (a single measurement)
  First meal (ad libitum breakfast) energy intake measurement. Participants will be served a standardised ad libitum breakfast in the laboratory. EI (kilocalories) will be measured objectively, by weighing foods before and after consumption and calculating energy intake based on their nutritional data.

SECONDARY OUTCOMES:
Palatability - Pleasantness | 9.5 hours: mean of ratings taken immediately following the three test meals and the two intakes of the test supplement (single measure), i.e., supplement, breakfast, lunch, supplement, dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used after each test meal: test supplement, breakfast, lunch, test supplement and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Filling | 9.5 hours: mean of ratings taken immediately following the three test meals and the two intakes of the test supplement (single measure), i.e., supplement, breakfast, lunch, supplement, dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used after each test meal: test supplement, breakfast, lunch, test supplement and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Satisfaction | 9.5 hours: mean of ratings taken immediately following the three test meals and the two intakes of the test supplement (single measure), i.e., supplement, breakfast, lunch, supplement, dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used after each test meal: test supplement, breakfast, lunch, test supplement and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Taste | 9.5 hours: mean of ratings taken immediately following the three test meals and the two intakes of the test supplement (single measure), i.e., supplement, breakfast, lunch, supplement, dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used after each test meal: test supplement, breakfast, lunch, test supplement and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Sweet | 9.5 hours: mean of ratings taken immediately following the three test meals and the two intakes of the test supplement (single measure), i.e., supplement, breakfast, lunch, supplement, dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used after each test meal: test supplement, breakfast, lunch, test supplement and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Palatability - Savoury | 9.5 hours: mean of ratings taken immediately following the three test meals and the two intakes of the test supplement (single measure), i.e., supplement, breakfast, lunch, supplement, dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used after each test meal: test supplement, breakfast, lunch, test supplement and dinner. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Pre-meal and changes in Composite Appetite Score | 9.5 hours: fast (pre-ONS), pre-breakfast: 90 (post-ONS), 60, 30 and 0 min; post-breakfast: 0 and 180 min (pre-lunch); post-lunch: 0 and 90 min (pre-ONS); 0 min post-ONS; estimated 120 min. post-ONS (pre-dinner); 0 min. post-dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at ten (10) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Composite Appetite Score is derived from VAS ratings of hunger, fullness, desire to eat and prospective food consumption. Fasting, mean and AUC values will be calculated.
Pre-meal and changes in Fullness | 9.5 hours: fast (pre-ONS), pre-breakfast: 90 (post-ONS), 60, 30 and 0 min; post-breakfast: 0 and 180 min (pre-lunch); post-lunch: 0 and 90 min (pre-ONS); 0 min post-ONS; estimated 120 min. post-ONS (pre-dinner); 0 min. post-dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at ten (10) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Fasting, mean and AUC values will be calculated.
Pre-meal and changes in Desire to Eat | 9.5 hours: fast (pre-ONS), pre-breakfast: 90 (post-ONS), 60, 30 and 0 min; post-breakfast: 0 and 180 min (pre-lunch); post-lunch: 0 and 90 min (pre-ONS); 0 min post-ONS; estimated 120 min. post-ONS (pre-dinner); 0 min. post-dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at ten (10) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Fasting, mean and AUC values will be calculated.
Pre-meal and changes in Prospective Food Consumption | 9.5 hours: fast (pre-ONS), pre-breakfast: 90 (post-ONS), 60, 30 and 0 min; post-breakfast: 0 and 180 min (pre-lunch); post-lunch: 0 and 90 min (pre-ONS); 0 min post-ONS; estimated 120 min. post-ONS (pre-dinner); 0 min. post-dinner
  Validated 100-millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, assessed at ten (10) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Fasting, mean and AUC values will be calculated.
Liking of test meals and supplements | Mean of ratings taken immediately following the three test meals and the two intakes of the test supplement (single measure), i.e., supplement, breakfast, lunch, supplement, dinner
  9-point likert scale from 0 dislike extremely to 9 like extremely
Pre-meal and changes in Glucose | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Insulin | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Growth Hormone | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Cortisol | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in GLP-1 | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in PYY | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Total Ghrelin | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Pre-meal and changes in Acylated Ghrelin | Up to 2 hours, from fast (morning) to immediately prior to breakfast meal: fasting (immediately before test supplement), and 30, 60, 90 minutes following ingestion of the test supplement
  Blood samples will be collected by a trained phlebotomist via cannula.
Total Energy intake (EI) (kilocalories) | 24 hours from breakfast, lunch and dinner meals, as well as from evening and night
  24-hour energy intake measurement derived from in-lab day trial plus free-living intake of standard meals plus food diary completed at home. Participants will be served a test supplement in two different time points, a standardised ad libitum breakfast, two standardised main meals (lunch and dinner) and will be required to complete a food diary from the dinner until bedtime. 24-hour EI (kilocalories) will be measured objectively, by weighing foods before and after consumption and calculating energy intake based on their nutritional data, and estimating caloric content from food diary provided. Total accumulated energy intake includes ad libitum breakfast meal, two test supplements, lunch meal, dinner meal and evening foods.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Leinster, Ireland